CLINICAL TRIAL: NCT05477849
Title: A Dose Escalation, Open-label Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Biologic Effect of VG2025 in the Treatment of Patients with Advanced Malignant Solid Tumors
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Biologic Effect of VG2025 in Patients with Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Virogin Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Virogin Biotech Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VG201-C101
Record Dates: First submitted 2022-07-15; First posted 2022-07-28 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Advanced Malignant Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 3+3 design (Experimental): This is an open label, single-arm trial using standard 3+3 design, in up to 30 HSV seropositive subjects. This rule-based design proceeds with cohorts of three patients
  Interventions: Drug: Recombinant Human IL12/15 Dual-Regulated Oncolytic HSV-1 Injection

INTERVENTIONS:
Drug: Recombinant Human IL12/15 Dual-Regulated Oncolytic HSV-1 Injection — 1. Dose level 1
  2. Dose level 2
  3. Dose level 3
  4. Dose level 4
  5. Dose level 5
  Other Names: VG2025

SUMMARY:
VG2025 is a Recombinant Human IL12/15 Dual-Regulated Oncolytic HSV-1 Injection. This Phase I study will be conducted in herpes simplex virus (HSV) -seropositive subjects with advanced malignant solid tumors that are refractory to conventional therapies. This is an open label study to determine the safety and tolerability of VG2025, and recommended dose of VG2025 for Phase II trials.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, dose-escalation trial using standard 3+3 dose-escalation design in patients with advanced malignant solid tumors. The trial will be conducted in multiple dosing cohorts, and evaluated for safety to determine the Maximum Tolerated Dose (MTD) and the Recommended Phase 2 Dose (RP2D). Dose limiting toxicity (DLT) evaluation period is for 4 weeks from the start of treatment Day 1 through Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent form.
2. Age 18 to 75 years (inclusive), male or female.
3. Subject with advanced malignant solid tumors who have failed standard treatment and for whom there is no effective treatment at this stage.
4. Eligible patients of childbearing potential (male and female) must agree to use a reliable method of contraception during the trial and for at least 90 days after dosing; females of childbearing potential must have a negative blood pregnancy test 7 days before enrollment.

Exclusion Criteria:

1. Subjects who have received other unlisted drugs clinical trial treatment 4 weeks before the first dose of the study drug.
2. Subjects who underwent major organ surgery (excluding needle biopsy) or had significant trauma 4 weeks before the first dose of the study drug.
3. In the herpes simplex virus recurrence and infection period, and there are corresponding clinical manifestations, such as oral herpes labialis, herpetic keratitis, herpetic dermatitis, genital herpes and so on.
4. Other active uncontrolled infection.
5. Known alcohol or drug dependence.
6. Subjects with mental disorders or poor compliance.
7. Women who are pregnant or breastfeeding.
8. Subjects in the opinion of the investigator are not suitable for this clinical study due to other serious systemic diseases or other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MTD/RP2D | During the 28 day DLT observation period
  Maximum tolerable dose (MTD) / Recommended dose for phase II (RP2D)
Adverse Events (AEs) and Serious Adverse Events (SAEs) | 12 months
  Occurence of Adverse Events (AEs) and Serious Adverse Events (SAEs)as assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0

SECONDARY OUTCOMES:
Level of deoxyribonucleic acid (DNA) | 12 months
  Shedding profile of detectable VG2025 deoxyribonucleic acid (DNA)
Interleukin level | 12 months
  Evaluate the interleukin-12 (IL-12) and interleukin-12 (IL-15) levels
ORR | Multiple time points before and after administration
  Objective response rate (ORR)
DCR | 12 months
  Disease control rate (DCR)
PFS | 12 months
  Progression-free survival (PFS)
OS | 12 months
  Overall Survival (OS)
Antibodies | 12 months
  VG2025 anti-drug antibodies (ADA) and neutralizing antibody (Nab)

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, M.D.，PhD, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital，Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No